CLINICAL TRIAL: NCT06463535
Title: Effects of Omega-3 as an Adjunct to Non-Surgical Periodontal Therapy on Chemerin Level
Brief Title: Effects of Omega-3 as an Adjunct to Non-Surgical Periodontal Therapy on Chemerin Level in Periodontitis Patients With Diabetes: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Ayman El-Gawish, lecturer, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BU7720
Record Dates: First submitted 2024-06-09; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus; Periodontal Diseases
MeSH Terms: conditions — Diabetes Mellitus; Periodontal Diseases | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group I (Experimental): Type 2 Diabetes Mellitus patients with CPD + SRP and Omega-3
  Interventions: Drug: Omega 3; Procedure: SRP alone
- group II (Active Comparator): Type 2 Diabetes Mellitus patients with CPD + SRP
  Interventions: Procedure: SRP alone

INTERVENTIONS:
Drug: Omega 3 — SRP + OMEGA 3
  Arms: group I
Procedure: SRP alone — Scaling and root planning

SUMMARY:
Patient grouping

* Group 1 (Type 2 Diabetes Mellitus patients with CPD + SRP and Omega-3)
* Group 2 (Type 2 Diabetes Mellitus patients with CPD + SRP) different clinical parameters were recorded ; plaque index (PI), gingival index (GI), probing depth (PD), and clinical attachment loss (CAL).

  6.Omega-3 poly-unsaturated fatty acids (1000mg) was given as an adjunctive treatment daily for 6 months to group 2, starting 2 weeks after phase 1 therapy.

DETAILED DESCRIPTION:
A parallel design randomized clinical trial was performed involving thirty participants divided into two groups, 15 participants in each group selected from the outpatient clinic in Oral medicine and Periodontology department.

Diabetic control was assessed by glycosylated hemoglobin A1c (HbA1c) of blood samples, patients had relatively stable glycemic control, as demonstrated by a difference not exceeding 1% in at least two HbA1c assays over the previous 6 m. HbA1c was assessed at baseline, 3m, and 6m.

Patient grouping

* Group 1 (Type 2 Diabetes Mellitus patients with CPD + SRP and Omega-3)
* Group 2 (Type 2 Diabetes Mellitus patients with CPD + SRP) Periodontal treatment protocol

Group 1 and 2 patients were treated by non-surgical approach in following steps:

1. Each patient had received an initial phase of detailed instruction in self-performed plaque control measures using soft toothbrush and interdental cleansing devices.
2. Full mouth SRP using ultrasonic scaler and hand instruments under local anesthesia was performed to each patient in two sessions.
3. Chlorehexidine CHX mouthwash was prescribed for patients to be used twice daily.
4. For each patient, follow up visits every 2 weeks were done to ensure plaque control.
5. Patients were re- examined after 2 weeks (baseline), 3 and 6 months

ELIGIBILITY:
Inclusion Criteria:

* Patients had type 2 DM for more than 2 years (diagnosed according to the American Diabetes Association criteria), with no other systemic problem. •Subjects had 14 or more natural teeth, of which at least five had a site with probing pocket depth (PPD) ≥ 5 mm and clinical attachment level ≥ 3 mm. From this point, according to the American Academy of Periodontology, subjects with moderate to severe periodontitis were included

Exclusion Criteria:

* Pregnant and breastfeeding women, smokers or former smokers, patients with other autoimmune or systemic disease, those patients who took antibiotics in the last 6 months and patients weren't willing to follow our study protocol or plaque regimen

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Serum level of chemerin | 6 months
  Serum level of chemerin

SECONDARY OUTCOMES:
periodontal clinical parameters | 6 months
  PD in mm
hba1c | 6 months
  Glycated Heamoglobin
GCF level of chemerin | 6 months
  GCF level of chemerin
periodontal clinical parameters | 6 months
  CAL in mm

CONTACTS AND LOCATIONS:
Locations (1):
- British University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ghalwash D, Ammar A, Hamdy A, El-Gawish A. Impact of the Adjunctive Use of Omega-3 in Periodontitis Patients With Diabetes on Local and Systemic Chemerin Levels: A Randomized Clinical Trial. Int J Dent. 2025 Jul 30;2025:7927250. doi: 10.1155/ijod/7927250. eCollection 2025. PMID 40771657